CLINICAL TRIAL: NCT00997880
Title: Effect of High-Dose and Low-Dose Statin for Coronary Plaque Modification
Brief Title: Statin and Atheroma Vulnerability Evaluation
Acronym: STABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, M.D., Ph.D.,Professor of Medicine Asan Medical Center, University of Ulsan, College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-0361
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease
Keywords: rosuvastatin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin calcium 40mg (Experimental): high-dose (40mg rosuvastatin)
  Interventions: Drug: Rosuvastatin calcium 40mg
- Rosuvastatin calcium10mg (Active Comparator): low-dose statin (10mg rosuvastatin)
  Interventions: Drug: Rosuvastatin calcium10mg

INTERVENTIONS:
Drug: Rosuvastatin calcium 40mg — Rosuvastatin calcium 40mg
  Other Names: CRESTOR® 40mg
  Arms: Rosuvastatin calcium 40mg
Drug: Rosuvastatin calcium10mg — Rosuvastatin 10mg
  Other Names: CRESTOR® 10mg
  Arms: Rosuvastatin calcium10mg

SUMMARY:
The purpose of this study is to evaluate the effect of statin therapy on the modification of atherosclerotic plaque composition and vulnerability in non-intervened coronary arteries with mild to moderate stenosis using VH-IVUS and OCT.

DETAILED DESCRIPTION:
At present, there is no proven drug or modality to stabilize the vulnerable plaques. A number of drugs that are beneficial for patients with coronary disease may act in part by improving the stability of plaques that are vulnerable for future rupture. Especially, Lipid-lowering therapy, particularly with statins, can stabilize vulnerable plaques or those that have already ruptured by improving endothelial function and reducing thrombogenicity, platelet aggregation, and possibly inflammation. As the atherosclerotic disease has progressed, there is an increase of the atherosclerotic plaque amounts. However, the changes of specific plaque compositions within the atherosclerotic lesions have not been sufficiently evaluated. Previous pathologic findings reported that there was a significant relation between the plaque size and necrotic core size.Conventional grey-scale intravascular ultrasound (IVUS) has significant limitations in accurately assessing atheromatous plaque composition. These limitations have been partially addressed by radiofrequency signal processing with spectral analysis of the back-scattered ultrasound signals. Using this technology, Virtual Histology (VH) IVUS is capable of characterizing plaque as calcified (white), fibrotic (dark-green), fibrofatty (yellow-green), and necrotic core (red). In addition, optical coherence tomography (OCT) is a light-based imaging modality that can be used in biological systems to study tissues in vivo with near-histologic, ultrahigh resolution. The rationale for intravascular application of OCT is its potential for in vivo visualizations of the coronary artery microstructure. This unique image resolution of OCT offers the potential to detect key features of vulnerable plaque in vivo. Beyond the inherent limitations of angioscopy and intravascular ultrasound, OCT might offer a much higher sensitivity in the detection of necrotic/lipid cores within coronary atheromas. Therefore, plaque characterization using VH-IVUS and OCT may provide detailed morphologic insights of plaque vulnerability.

We hypothesized that statin would provide benefits to stabilize coronary plaque composition by LDL-reduction and/or a pleiotropic effect. We also hypothesized that high-dose statin would be more beneficial in reducing the vulnerable plaque and stabilizing the vulnerable plaque composition than low-dose statin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age inclusive.
2. Patients with stable (CCS class 1 to 4) or acute coronary syndromes (unstable angina pectoris Braunwald class IB, IC, IIB, IIC, IIIB, IIIC or NSTEMI) or patients with atypical chest pain or without symptoms but having documented myocardial ischemia who will undergo either planned coronary angiography, or percutaneous coronary intervention
3. Non-culprit de novo lesion in a native coronary artery with at least one deferred coronary lesion with 1) visually-estimated angiographic % diameter stenosis 20-50% or 2) % diameter stenosis >50% without any evidence of inducible ischemia (FFR≥0.8 or negative perfusion on thiallium scan or negative treadmill test). Index lesion should have at least 1 fibroatheroma or TCFA.
4. The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site

Exclusion Criteria:

1. Planned cardiac surgery (e.g., CABG, valve repair or replacement, or aneurysmectomy) or planned major non-cardiac surgery within the study period
2. Stroke or resuscitated sudden death in the past 6 months
3. Chronic disease requiring treatment with oral, intravenous, or intra-articular corticosteroids (use of topical, inhaled, or nasal corticosteroids is permissible)
4. Untreated hyperthyroidism, or hypothyroidism with TSH levels more than 1.5 times upper limit of normal
5. A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer
6. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study
7. Evidence of congestive heart failure, or left ventricular ejection fraction < 40%
8. Significant renal disease manifested by serum creatinine > 2.0mg/dL, or creatinine clearance of < 40 ml/min (by Cockcroft-Gault method)
9. Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal)
10. History of myopathy or elevated creatine kinase (CK) > 3 times upper normal limit at screening
11. History of adult asthma manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s)
12. Unwillingness or inability to comply with the procedures described in this protocol
13. History of any arterial bypass or angioplastic intervention involving the target vessel
14. The luminal narrowing in the target vessel or in the left main coronary artery >50% by visual inspection of angiogram
15. Luminal diameter of the target vessel < 2.5mm by visual inspection of coronary angiogram
16. Presence of thrombus or complex plaque morphology in the target vessel that suggests a high likelihood of distal embolism
17. Severe tortuosity of the target vessel or any other anatomical reasons that the investigator deems inappropriate for IVUS procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent compositional change of coronary plaque in the entire pullback length Percent compositional c Percent hange of coronary plaque in the entire pullback length of "target segment" (within both proximal and distal fiduciary sites) | 12months

SECONDARY OUTCOMES:
VH-IVUS parameters | 12months
Conventional IVUS parameters | 12months
OCT Sub-study parameters | 12months
Serum biomarkers | 12months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD,PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (1):
- Asan Medical Center, Seoul, Republic of Korea, South Korea

REFERENCES:
- [Derived] Kwon O, Kang SJ, Kang SH, Lee PH, Yun SC, Ahn JM, Park DW, Lee SW, Kim YH, Lee CW, Han KH, Park SW, Park SJ. Relationship Between Serum Inflammatory Marker Levels and the Dynamic Changes in Coronary Plaque Characteristics After Statin Therapy. Circ Cardiovasc Imaging. 2017 Jul;10(7):e005934. doi: 10.1161/CIRCIMAGING.116.005934. PMID 28679524
- [Derived] Park SJ, Kang SJ, Ahn JM, Chang M, Yun SC, Roh JH, Lee PH, Park HW, Yoon SH, Park DW, Lee SW, Kim YH, Lee CW, Mintz GS, Han KH, Park SW. Effect of Statin Treatment on Modifying Plaque Composition: A Double-Blind, Randomized Study. J Am Coll Cardiol. 2016 Apr 19;67(15):1772-1783. doi: 10.1016/j.jacc.2016.02.014. PMID 27081016